CLINICAL TRIAL: NCT05610826
Title: Preoperative PRRT Versus Surgical Cytoreduction Alone in Metastatic Pancreatic Neuroendocrine Tumors to the Liver: A Phase II Multi-institutional Trial
Brief Title: Preoperative PRRT Versus Surgical Cytoreduction in Metastatic Pancreatic Neuroendocrine Tumors to the Liver
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: 0 enrollment
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-1485
Record Dates: First submitted 2022-11-02; First posted 2022-11-09 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Neuroendocrine Tumor; Pancreas Cancer
Keywords: pancreatic cancer; pancreas cancer
MeSH Terms: conditions — Adenoma, Islet Cell; Pancreatic Neoplasms | interventions — Cytoreduction Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1- Control Arm - Standard Of Care - no peptide receptor radionuclide therapy (Other): Arm 1 is the control arm, which will undergo standard of care cytoreductive surgery (for the tumor). Participants in this arm will not receive peptide receptor radionuclide therapy (PRRT).
  Interventions: Procedure: cytoreductive surgery
- Arm 2 (peptide receptor radionuclide therapy + cytoreductive surgery) (Experimental): Arm 2 will undergo four cycles of peptide receptor radionuclide therapy (PRRT) before cytoreductive surgery.
  Interventions: Procedure: cytoreductive surgery; Drug: Lutathera - a small molecule used in Peptide Receptor Radionuclide Therapy (PRRT); Procedure: Peptide receptor radionuclide therapy (PRRT)

INTERVENTIONS:
Procedure: cytoreductive surgery — Cytoreductive surgery is an operation to remove as much tumor tissue as possible.
Drug: Lutathera - a small molecule used in Peptide Receptor Radionuclide Therapy (PRRT) — PRRT is a form of targeted treatment (think of a "lock and key") done by the use of a small molecule (Lutathera). Lutathera acts as a "key" to "lock" onto certain areas your tumor cells called receptors when injected into a vein and travels through blood.
  Arms: Arm 2 (peptide receptor radionuclide therapy + cytoreductive surgery)
Procedure: Peptide receptor radionuclide therapy (PRRT) — PRRT is a molecular targeted therapy used to treat neuroendocrine tumors (NET). Molecular targeted therapies use drugs or other substances to identify and attack cancer cells while reducing harm to healthy tissue. PRRT delivers high doses of radiation to tumors in the body to destroy or slow their growth and reduce disease side effects.
  Arms: Arm 2 (peptide receptor radionuclide therapy + cytoreductive surgery)

SUMMARY:
Doctors and researchers leading this study hope to learn more about peptide receptor radionuclide therapy (PRRT) in combination with cytoreduction (surgically removing tumors). They hope to learn if combining PRRT in combination with cytoreduction would be more effective than cytoreduction alone. PRRT itself is approved by the U.S. Food and Drug Administration (FDA) for people with PanNETs however the combination with cytoreduction is considered experimental.

Your participation in this research will last about 2 years. The purpose of this research is to gather information on the safety and effectiveness of PRRT.

DETAILED DESCRIPTION:
Doctors and researchers leading this study hope to learn more about peptide receptor radionuclide therapy (PRRT) in combination with cytoreduction (surgically removing tumors). They hope to learn if combining PRRT in combination with cytoreduction would be more effective than cytoreduction alone. PRRT itself is approved by the U.S. Food and Drug Administration (FDA) for people with PanNETs however the combination with cytoreduction is considered experimental.

Your participation in this research will last about 2 years. The purpose of this research is to gather information on the safety and effectiveness of PRRT.

PRRT is a form of targeted treatment (think of a "lock and key") done by the use of a small molecule (Lutathera) Lutathera acts as a "key" to "lock" onto certain areas your tumor cells called receptors when injected into a vein and travels through the bloodstream. Lutetium-177 is the radionuclide in Lutathera which is a chemical that delivers strong radiation directly into your tumor cells and works by causing death of the cancerous tissues.

PRRT can only be done on patients who have tumors that have the somatostatin receptors. Before being given PRRT, your treating doctor will run imaging tests to make sure your tumors have these targeted receptors. Your participation in this research will last about 2 years. The purpose of this research is to gather information on the safety and effectiveness of PRRT.

Participants will be randomized (like the flip of a coin) to one of two arms. Arm 1 is the control arm, which will undergo standard of care cytoreductive surgery (for the tumor). Arm 2 will undergo four cycles of PRRT before cytoreductive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic Pancreatic neuroendocrine tumors (PanNET) to the liver
* Well- or moderately differentiated (grade 1 or grade 2, Ki-
* Ability to aim for equal or greater than 90% hepatic cytoreduction surgically
* Proof of SSTR2 expression by uptake of tumor on 68Ga DOTATATE PET CT (Krenning Score on all or a majority of lesions
* Age older than 18 years
* No Somatostatin Analogues (SSA) or other systemic therapy for 4 weeks prior to starting PRRT, if randomized to arm 2.

Exclusion Criteria:

* Patient with G3 or poorly differentiated NET (grade 3, Ki-67 >20%)
* Previous liver-directed therapy with Yttrium-90 (TACE/TAE allowed if performed more than 12 months prior to enrollment)
* Systemic therapy with Capecitabine and/or Temozolamide within 12 months of enrollment.
* No tumor uptake on 68Ga DOTATATE PET CT
* Liver tumor burden > 50% (as defined by CT or MRI)
* Signs of early liver failure (T-Bilirubin >3, INR > 1.5, Albumin <3.0 g/dL unless prothrombin time is within the normal range) or cirrhosis or ascites
* calculated by the Cockroft Gault method, eventually confirmed by measured creatinine clearance
* (or measured glomerular filtration rate (GFR) using plasma clearance methods, not gamma
* camera-based) <50 mL/min (the measured creatinine clearance / GFR is required only as - confirmatory exam).
* 2. Hb concentration <5.0 mmol/L (<8.0 g/dL); WBC <2x109/L (2000/mm3); platelets <75x109/L - (75x103/mm3).
* Known brain metastases, unless these metastases have been treated and stabilized.
* Uncontrolled congestive heart failure (NYHA II, III, IV).
* Uncontrolled diabetes mellitus as defined by a fasting blood glucose >2 ULN.
* Pregnancy or lactation.
* For female patients of childbearing potential (defined as < 2 years after last menstruation and not surgically sterile) and male patients, who are not surgically sterile or with female partners of childbearing potential: absence of effective, non-hormonal means of contraception (intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal gel). - Prior external beam radiation therapy to more than 25% of the bone marrow.
* Current spontaneous urinary incontinence making impossible the safe administration of the radioactive IMP.
* Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and with no evidence of recurrence.
* Patients who have not provided a signed informed consent form to accept this treatment.
* Poor renal function
* Quality Unit language added
* editorial changes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival | 2 years
  To determine whether preoperative peptide receptor radionuclide therapy (PRRT) prior to hepatic cytoreduction increases progression free survival (PFS1) (when compared to cytoreduction alone) in patients with metastatic PanNETs to the liver

SECONDARY OUTCOMES:
Overall Survival | 2 years
  To determine whether preoperative peptide receptor radionuclide therapy (PRRT) prior to hepatic cytoreduction increases overall survival.
  (when compared to cytoreduction alone) in patients with metastatic PanNETs to the liver
Objective Response Rate | 2 Years
  To determine whether preoperative peptide receptor radionuclide therapy (PRRT) induces a significant objective response rate (according to RECIST) in the primary tumor (if available) and hepatic metastases of patients with metastatic PanNETs to the liver, thus facilitating surgical resection.
Increase in Progression Free Survival | 2 years
  To determine whether PRRT plus cytoreductive surgery increases PFS when compared to a historical cohort of patients undergoing PRRT only for metastatic PanNETs.
Improvement in Progression-Free Survival (PFS2) | 2 years
  To determine whether PRRT plus cytoreduction compared to cytoreduction alone followed by PRRT once progression has occurred improves progression-free survival (PFS2)
Improvement in Overall Survival | 2 years
  To determine whether PRRT plus cytoreduction compared to cytoreduction alone followed by PRRT once progression has occurred improves Overall Survival.
Difference in imaging characteristics | 2 years
  To determine differences in imaging characteristics (e.g. tumor size), biochemical and molecular signatures of patients having received surgery + PRRT or surgery alone.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Keutgen, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States